CLINICAL TRIAL: NCT06692166
Title: A Randomized, Open-label, Phase 3 Study to Evaluate 9MW2821 vs Treatment of Physician's Choice in Subjects With Recurrent or Metastatic Cervical Cancer Who Progressed on or After Platinum-based Chemotherapy
Brief Title: A Study to Evaluate 9MW2821 Versus Treatment of Physician's Choice for Subjects With Recurrent or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-CP304
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Cervical Cancer
Keywords: Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Uterine Cervical Diseases; Uterine Diseases; Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Uterine Cervical Diseases; Uterine Diseases | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW2821 (Experimental)
  Interventions: Drug: 9MW2821
- Treatment of Physician's Choice (Active Comparator)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: 9MW2821 — 1.25mg/kg of 9MW2821 by intravenous infusion on days 1, 8 and 15 of every 28-day cycle
  Arms: 9MW2821
Drug: Chemotherapy — 1.0 or 1.25 mg/m ^2 topotecan by intravenous infusion on days 1 to 5 or 1000 mg/m ^2 gemcitabine by intravenous infusion on days 1 and 8 or 500 mg/m ^2 pemetrexed by intravenous infusion on day 1 of every 21 days
  Arms: Treatment of Physician's Choice

SUMMARY:
The purpose of this study is to compare the efficacy and safety of 9MW2821 and chemotherapy in participants with recurrent or metastatic cervical cancer who progressed on or after platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form.
2. Female subjects aged 18 to 75 years (including 18 and 75 years).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed recurrent or metastatic cervical cancer (squamous cell, HPV-associated adenocarcinoma, or adenosquamous), not amenable to resection or chemoradiation with curative intent.
5. Subject must have received a platinum-based chemotherapy with or without bevacizumab and received no more than 2 prior systemic therapy in the metastatic/recurrent setting. Subject must have experienced radiographic progression during or after the last treatment regimen.
6. An archival tumor tissue sample or a fresh tissue sample should be provided.
7. Life expectancy of ≥ 12 weeks.
8. Subjects must have measurable disease according to RECIST (version 1.1).
9. Adequate to receive one of the chemotherapy regimens in the control group (gemcitabine, pemetrexed, topotecan);
10. Adequate organ functions.
11. Sexually active fertile subjects must agree to use methods of contraception during the study and at least 6 months after termination of study therapy.
12. Subjects are willing to follow study procedures.

Exclusion Criteria:

1. Has other histologies not mentioned as part of the inclusion criteria above, i.e. HPV-independent adenocarcinoma or primary neuroendocrine.
2. Chemotherapy or radiotherapy within 21 days prior to the first dose of study drug, traditional Chinese medicine with anticancer indication within 14 days prior to the first dose of study drug, use of any investigational drug or device within 28 days prior to the first dose of study drug, received treatment of nectin-4 targeted ADC, received treatment of ADC with MMAE payload, received any strong CYP3A4 inhibitors within 14 days prior to the first dose of study drug.
3. Preexisting treatment related toxicity Grade ≥ 2. Subjects experienced Grade ≥ 3 immune related adverse events during or after immunotherapy.
4. Subjects had clinically significant hydronephrosis that could not be relieved by nephrostomy or urethral stenting, as determined by the investigator.
5. Major surgery within 28 days prior to first dose of study drug.
6. Hemoglobin A1C (HbA1c) ≥ 8%.
7. Preexisting peripheral neuropathy Grade ≥ 2.
8. Any live vaccines within 28 days before first dose of study drug or during the study.
9. Documented history of clinically significant cardiac or cerebrovascular diseases within 6 months prior to the first dose of study drug.
10. Other severe or uncontrolled disease, i.e. severe respiratory system disease, thromboembolic events, active bleeding or active infection.
11. Central nervous system metastases.
12. History of another malignancy within 3 years before the first dose of study drug. Subjects with cured malignancies are allowed.
13. History of autoimmune disease requiring systemic treatment within 2 years before the first dose of study drug.
14. Has ocular conditions that may increase the risk of corneal epithelium damage.
15. Known sensitivity to any of the ingredients of the investigational product; History of drug abuse or mental illness.
16. Uncontrolled tumor-related bone pain or spinal cord compression.
17. Pleural effusion, ascites or pericardial effusion with syptoms or needed drainage.
18. Condition or situation which may put the subject at significant risk.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-12-09 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 3 years
  Time from the date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate per investigator | Up to 3 years
  The percentage of subjects who experience a best response of either CR or PR.
Disease Control Rate per investigator | Up to 3 years
  The percentage of subjects who experience a best response of CR, PR or stable disease (SD).
Progression Free Survival per investigator | Up to 3 years
  Time from the date of first randomization to the earliest date of documented disease progression per radiological evidence or death from any cause.
Duration of Response per investigator | Up to 3 years
  Time from the date of the first complete response (CR) or partial response (PR) to the earliest date of disease progression or death from any cause.
Time to response per investigator | Up to 3 years
  Time from the date of randomization to the date of CR or PR.
Incidence of adverse events | Up to 3 years
Incidence of Anti-Drug Antibody (ADA) | Up to 3 years

OTHER OUTCOMES:
Mean change from baseline in the European Organisation for Research and Treatment of Cancer (EORTC) 30-item core quality-of-life questionnaire (QLQ-C30） | Up to 3 years
  The EORTC QLQ-C30 is a 30-question instrument designed to assess overall QoL in cancer patients with 15 domains: 1 GHS/QoL scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptomatic scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). Most items were scored from 1 ("not at all") to 4 ("very much"), with the exception of items contributing to the GHS/QoL, which were scored from 1 ("very poor") to 7 ("excellent"). Raw scores were linearly transformed so that all transformed scores ranged from 0 to 100. For the overall health status/quality of life scale and the 5 functioning scales, high scores indicated better overall health status/functioning, and negative change from baseline indicated less improvement. For the symptom scales, a high score indicates a high level of symptomatology, while a negative change from baseline indicates improvement in symptoms.
EORTC Quality of Life Questionnaire Cervical Cancer Module (QLQ-CX24) Total Scores | Up to 3 years
  The EORTC QLQ-CX24 questionnaire is intended for patients with cervical cancer with different disease stages and treatment modalities. The EORTC-QLQ-CX24 questionnaire consists of 24 questions with answers ranging from 1 (not at all) to 4 (very much). Four functional scales and five symptom scales will be calculated using the EORTC QLQ-CX24 Scoring Manual. The 9 scores calculated from the EORTC-QLQ-CX24 questionnaire will be summarized in descriptive statistics by treatment arm. A high score indicates a high level of symptomatology, while a negative change from baseline indicates improvement in symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Liu R, Wang S, Feng Z, Yang H, Gao S, Li X, Yao X, Chen J, Gong Z, Li Y, Li X, Wang S, Hu C, Liu J, Zhang M, Yuan F, Shi B, Lou H, Zhao P, Qiu F, Guo H, Hu B, Xu D, Huang H, Zhang X, Feng M, Wang X, Li G, Liu D, Chen X, Wang P. Bulumtatug Fuvedotin (BFv, 9MW2821), a next-generation Nectin-4 targeting antibody-drug conjugate, in patients with advanced solid tumors: a first-in-human, open-label, multicenter, phase I/II study. Ann Oncol. 2025 Aug;36(8):934-943. doi: 10.1016/j.annonc.2025.04.009. Epub 2025 Apr 25. PMID 40288679